CLINICAL TRIAL: NCT05688852
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of VTX958 in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: VTX958 for the Treatment of Moderately to Severely Active Crohn's Disease
Acronym: Harmony-CD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Ventyx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTX958-202
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease
Keywords: VTX958; Harmony; Crohn's disease; TYK2
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will employ a double-blind design. Participants, Investigators, study center staff, persons performing the assessments, and the Sponsor are to remain blinded to the identity of the Induction and Maintenance Period treatment from the time of randomization until the interim database lock for the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VTX958 Dose A (Experimental)
  Interventions: Drug: VTX958
- VTX958 Dose B (Experimental)
  Interventions: Drug: VTX958
- VTX958 Placebo (Placebo Comparator)
  Interventions: Drug: VTX958 Placebo

INTERVENTIONS:
Drug: VTX958 — Dose A VTX958
  Arms: VTX958 Dose A
Drug: VTX958 — Dose B VTX958
  Arms: VTX958 Dose B
Drug: VTX958 Placebo — Placebo
  Arms: VTX958 Placebo

SUMMARY:
This is a multicenter, randomized, double-blind placebo-controlled, parallel group study to evaluate the efficacy and safety of VTX958 in participants with moderately to severely active Crohn's Disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind placebo-controlled, parallel group study to evaluate the efficacy and safety of VTX958 in participants with moderately to severely active Crohn's Disease. Approximately 93 eligible patients will be randomized, and randomization will be stratified by prior use of biologics for the treatment of CD (yes/no).

The study consists of a 30-day Screening Period, a 12-week double-blind Induction Treatment Period, a 40-week double-blind Maintenance Treatment Period, an Open-Label Extension (OLE) of up to 144 weeks, and a 30-day safety Follow-Up Period. The maximum duration of treatment will be 36 months, including the Induction, Maintenance, and OLE Periods. For all participants, a Follow-Up visit will be performed at 30 days after the last dose of study drug.

Objectives Primary Objectives

* Evaluate the efficacy of VTX958 in achieving reduction in Crohn's Disease Activity Index (CDAI) score at the end of the Induction Period

Secondary Objectives

* Evaluate the efficacy of VTX958 in inducing clinical and symptomatic response and remission at the end of the Induction Period
* Evaluate the efficacy of VTX958 in inducing endoscopic response and clinical remission at the end of the Induction Period

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 18 to 75 years of age, inclusive, at the time of consent
2. Capable of giving signed informed consent
3. Documented diagnosis of CD ≥ 3 months prior to Day 1. The diagnosis of CD must be confirmed by clinical, endoscopic, and histologic evidence.
4. Moderately to severely active CD

Exclusion Criteria:

1. Current diagnosis of ulcerative colitis, indeterminate colitis, microscopic colitis, ischemic colitis, or infectious colitis
2. Presence of a stoma or ileoanal pouch
3. Presence of currently known complications of CD such as symptomatic bowel stricture(s) and >2 missing segments of the following 5 segments: terminal ileum, right colon, transverse colon, left and sigmoid colon, and rectum, fulminant colitis, toxic megacolon or any other manifestation that may require surgery or hospitalization
4. Known diagnosis of short gut or bowel syndrome
5. Previous exposure to VTX958 or any other TYK2 inhibitor (eg, deucravacitinib) in any study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in mean Crohn's disease Activity Index (CDAI) score from baseline to week 12 | During screening to week 12
  Change in Mean CDAI (Crohn's disease Activity Index). CDAI is a weighted index comprising eight Crohn's Disease (CD)-related clinical and laboratory variables, to assess CD disease activity. Three of the variables, stool frequency, abdominal pain, and general well-being, are patient-reported measures recorded daily. The total CDAI score is calculated using the sum of each variable times the multiplier. The total score range of the CDAI is from 0 to 600.

SECONDARY OUTCOMES:
The proportion of participants achieving endoscopic response at Week 12 | During screening to week 12
  SES-CD is an endoscopic grading system is used to assess CD disease activity. The SES-CD assesses 4 endoscopic variables: the size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each variable score ranging from 0 to 3. The total SES-CD score is calculated using the sum of all parameter scores in 5 segments: terminal ileum, right colon, transverse colon, left colon, and rectum.
Change from baseline in mean simple endoscopic score in Crohn's disease SES-CD at Week 12 | During screening to week 12
  Change from baseline in mean simple endoscopic score in Crohn's disease SED-CD at 12 weeks. The SES-CD is an endoscopic grading system is used to assess CD disease activity. The SES-CD assesses 4 endoscopic variables: the size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each variable score ranging from 0 to 3. The total SES-CD score is calculated using the sum of all parameter scores in 5 segments: terminal ileum, right colon, transverse colon, left colon, and rectum.
Proportion of participants achieving clinical remission at Week 12 | During screening to week 12
  Clinical remission is defined as a CDAI score < 150. CDAI is a weighted index comprising eight Crohn's Disease (CD)-related clinical and laboratory variables, to assess CD disease activity. Three of the variables, stool frequency, abdominal pain, and general well-being, are patient-reported measures recorded daily. The total CDAI score is calculated using the sum of each variable times the multiplier. The total score range of the CDAI is from 0 to 600.
Proportion of participants achieving patient-reported outcome 2 (PRO2) remission at Week 12 | During screening to week 12
  The proportion of participants achieving PRO2 remission at week 12. PRO2 remission is defined is an unweighted CDAI component of daily AP score ≤ 1 and unweighted CDAI component of daily average stool frequency (SF) score ≤ 3
Proportion of participants achieving clinical response at Week 12 | During screening to week 12
  Proportion of participants achieving clinical response at Week 12. A clinical response is defined as ≥ 100 points reduction from baseline in CDAI score or CDAI score < 150. CDAI is a weighted index comprising eight Crohn's Disease (CD)-related clinical and laboratory variables, to assess CD disease activity. Three of the variables, stool frequency, abdominal pain, and general well-being, are patient-reported measures recorded daily. The total CDAI score is calculated using the sum of each variable times the multiplier. The total score range of the CDAI is from 0 to 600.
Proportion of participants achieving both endoscopic response (outcome- measure # 2) and clinical remission (outcome measure # 4) at Week 12 | During screening to week 12
  Proportion of participants achieving both endoscopic response (as described in outcome measure 2) and clinical remission (as described in outcome measure 4) at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Naik, PhD, Study Director — Ventyx Biosciences, Inc
Locations (105):
- United States (26):
  - Local Site # 840105, Garden Grove, California
  - Local Site # 840109, Lancaster, California
  - Local Site # 840124, Kissimmee, Florida
  - Local Site # 840104, Miami, Florida
  - Local Site # 840108, Orlando, Florida
  - Local Site # 840125, Orlando, Florida
  - Local Site # 840112, Atlanta, Georgia
  - Local Site # 840115, Glenview, Illinois
  - Local Site # 840107, Gurnee, Illinois
  - Local Site # 840119, New Albany, Indiana
  - Local Site # 840127, Louisville, Kentucky
  - Local Site # 840113, Shreveport, Louisiana
  - Local Site # 840117, Chevy Chase, Maryland
  - Local Site # 840118, Rockville, Maryland
  - Local Site # 840116, Liberty, Missouri
  - Local Site # 840121, Winston-Salem, North Carolina
  - Local Site # 840122, Columbus, Ohio
  - Local Site # 840106, Oklahoma City, Oklahoma
  - Local Site # 840123, Myrtle Beach, South Carolina
  - Local Site # 840111, Garland, Texas
  - Local Site # 840103, Katy, Texas
  - Local Site # 840110, Lubbock, Texas
  - Local Site # 840114, Lubbock, Texas
  - Local Site # 840102, Southlake, Texas
  - Local Site # 840101, Tyler, Texas
  - Local Site # 840126, West Jordan, Utah
- Australia (6):
  - Local Site # 036106, Concord
  - Local Site # 036103, Melbourne
  - Local Site # 036104, Melbourne
  - Local Site # 036101, Melbourne
  - Local Site # 036102, Parkville
  - Local Site # 036105, Perth
- Brazil (7):
  - Local Site # 076102, Taguatinga, Federal District
  - Local Site # 076104, Porto Alegre, Rio Grande Do Su
  - Local Site # 076106, Curitiba
  - Local Site # 076107, Curitiba
  - Local Site # 076101, Santo André
  - Local Site # 076103, São Paulo
  - Local Site # 076105, São Paulo
- Bulgaria (3):
  - Local Site # 100102, Rousse
  - Local Site # 100103, Sofia
  - Local Site # 100101, Sofia
- Canada (4):
  - Local Site # 124103, Oakville, Ontario
  - Local Site # 124104, Oshawa, Ontario
  - Local Site # 124101, Toronto, Ontario
  - Local Site # 124102, Woodbridge, Ontario
- Czechia (6):
  - Local Site # 203106, Brno
  - Local Site # 203102, Brno
  - Local Site # 203105, Hradec Králové
  - Local Site # 203104, Ostrava
  - Local Site # 203101, Slaný
  - Local Site # 203103, Ústí nad Labem
- Georgia (3):
  - Local Site # 268105, Tbilisi
  - Local Site # 268103, Tbilisi
  - Local Site # 268101, Tbilisi
- Germany (7):
  - Local Site # 276102, Tübingen, Baden-Wurttemberg
  - Local Site # 276105, Ulm, Baden-Wurttemberg
  - Local Site # 276106, Duisburg, North Rhine-Westphalia
  - Local Site # 276109, Berlin
  - Local Site # 276104, Berlin
  - Local Site # 276108, Hessen
  - Local Site # 276107, Kiel
- Hungary (6):
  - Local Site # 348102, Békéscsaba
  - Local Site # 348101, Budapest
  - Local Site # 348106, Gyöngyös
  - Local Site #348104, Szeged
  - Local Site # 348103, Szekszárd
  - Local Site # 348105, Tatabánya
- Israel (6):
  - Local Site # 376103, Ashkelon
  - Local Site # 376108, Haifa
  - Local Site # 376105, Jerusalem
  - Local Site # 376107, Jerusalem
  - Local Site # 376101, Petah Tikva
  - Local Site # 376102, Rehovot
- Italy (6):
  - Local Site # 380104, Milan, Lombardy
  - Local Site # 380105, Negrar, Verona
  - Local Site # 380101, Bari
  - Local Site # 380107, Milan
  - Local Site # 380109, Rome
  - Local Site # 380106, Turin
- Local Site # 440101, Vilnius, Lithuania
- Moldova (2):
  - Local Site # 498101, Chisinau
  - Local Site # 498102, Chisinau
- Poland (17):
  - Local Site # 616116, Bydgoszcz
  - Local Site #616113, Knurów
  - Local Site # 616112, Krakow
  - Local Site # 616110, Lodz
  - Local Site # 616105, Lodz
  - Local Site # 616101, Lodz
  - Local Site # 616117, Lublin
  - Local Site # 616109, Nowy Targ
  - Local Site # 616107, Oświęcim
  - Local Site # 616115, Poznan
  - Local Site # 616104, Rzeszów
  - Local Site # 616118, Staszów
  - Local Site # 616106, Szczecin
  - Local Site # 616102, Warsaw
  - Local Site # 616114, Wroclaw
  - Local Site # 616103, Wroclaw
  - Local Site # 616108, Wroclaw
- Slovakia (5):
  - Local Site # 703103, Bratislava
  - Locla Site # 703101, Košice
  - Local Site # 703106, Martin
  - Local Site # 703104, Prešov
  - Local Site # 703102, Šahy

IPD SHARING:
Plan to Share IPD: Undecided